CLINICAL TRIAL: NCT05245682
Title: Early-Phase Open-label Study of Tolinapant and Radiation in Cisplatin-Ineligible Patients With Previously Untreated, Locally Advanced Head and Neck Cancer
Brief Title: Tolinapant and Radiation for Cisplatin-Ineligible, Previously Untreated, Locally Advanced Head and Neck Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nicole Schmitt, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002992; P30CA138292 (NIH); WINSHIP5380-21 (Other: Emory University); NCI-2021-09678 (Registry Identifier: CTRP)
Record Dates: First submitted 2022-01-11; First posted 2022-02-18 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Carcinoma of Unknown Primary; Locally Advanced Head and Neck Squamous Cell Carcinoma; Locally Advanced Hypopharyngeal Squamous Cell Carcinoma; Locally Advanced Laryngeal Squamous Cell Carcinoma; Locally Advanced Nasopharyngeal Squamous Cell Carcinoma; Locally Advanced Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: interventions — ASTX-660; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (tolinapant, radiation therapy) (Experimental): Patients undergo standard of care radiation therapy for a total of 35 fractions over 7 weeks and receive tolinapant PO daily for 7 days during weeks 1, 3, 5, and 7 of radiation therapy in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Tolinapant; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Tolinapant — Given PO
  Other Names: ASTX660; 1799328-86-1; XIAP/cIAP1 Antagonist ASTX660
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT Therapy

SUMMARY:
This early-phase trial tests the safety and side effects of a tolinapant given together with radiation therapy in treating patients with head and neck cancer for which the patient has not received treatment in the past (previously untreated), has spread to nearby tissue or lymph nodes (locally advanced) and cannot receive cisplatin (cisplatin-ineligible). Tolinapant may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving tolinapant and radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the safety and tolerability of the recommended phase 2 dose (RP2D) of tolinapant when given in combination with radiation.

Secondary Objectives:

To assess preliminary efficacy of the combination of tolinapant and radiation in cisplatin ineligible patients with head and neck cancer as determined by locoregional control, two year progression-free survival (PFS), and two-year overall survival (OS).

Exploratory Objective:

To compare immune cell infiltrates following the first cycle of tolinapant + radiation, compared with baseline biopsy tissue and peripheral blood.

TERTIARY/EXPLORATORY OBJECTIVES:

I. To assess the effects of the combination of tolinapant + radiation on immune cells in blood and tumor.

II. To assess the association between immune responses and FADD expression in tumors.

OUTLINE:

Patients undergo standard of care radiation therapy for a total of 35 fractions over 6-7 weeks and receive tolinapant orally (PO) daily for 7 days during weeks 1, 3, 5, and 7 of radiation therapy in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up 1, 3, 6, 12, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female.
2. Age ≥18 years.
3. ECOG performance status ≤1 (see Appendix A).
4. Patients with histologically or cytologically confirmed diagnosis of HNSCC, previously untreated and locally advanced, for whom definitive or adjuvant radiation is planned but cisplatin chemotherapy is contraindicated.

   For the purposes of trial eligibility, anatomic subsites of HNSCC may include the larynx, oropharynx, hypopharynx, nasopharynx, or unknown primary site presenting with neck lymph nodal disease.

   Patients must have a contraindication to cisplatin as defined below. The scores must be recorded on a CRF:

   Age ≥ 70 with moderate to severe comorbidity, defined as having one or more of the following conditions within 30 days prior to registration:
   * Modified Charlson Comorbidity Index ≥ 1
   * ACE-27 Index ≥ 1
   * G-8 score ≤ 14
   * CARG Toxicity Score ≥ 30%
   * CIRS-G Score ≥ 4 -OR-

   Age ≥ 18 with an absolute or relative contraindication to cisplatin, defined as one or more of the following criterion within 30 days prior to registration:
   * Pre-existing peripheral neuropathy grade ≥ 1;
   * History of hearing loss, defined as either an existing need of a hearing aid OR moderate hearing loss as defined by the American Speech and Hearing Association (pretreatment audiogram showing 40-55 db HL hearing loss)
   * Creatinine clearance (CrCl) must be > 30 and < 50 mL/min. For this calculation, use the Cockroft-Gault formula: CrCl = 0.85 (if female)* ((140-Age) / (Serum Creatinine)) * (Weight in kg / 72).
5. Acceptable organ function, as evidenced by the following laboratory data:

   * Absolute neutrophil count [ANC] ≥ 1,500 cells/l; hemoglobin ≥ 9 g/dl, platelets ≥ 100,000/l.
   * Serum creatinine ≤ 1.5 mg/dl, or calculated creatinine clearance ≥ 60 ml/min.
   * Bilirubin ≤ upper limit normal [ULN], alanine aminotransferase [ALT] ≤ 1.5 x ULN and/or aspartate aminotransferase [AST] ≤ 1.5 x ULN, alkaline phosphatase ≤ 2.5 x ULN.
   * Prothrombin time (PT)/international normalized ratio (INR) ≤ 1.5 x ULN.
   * Activated partial thromboplastin (aPTT) time ≤ 1.5 x ULN. Amylase and lipase ≤ ULN.
6. The effects of tolinapant on the developing human fetus are unknown. For this reason and because tolinapant as well as other therapeutic agents used in this trial are known to be teratogenic, females of child-bearing potential (FCBP) must have a negative serum pregnancy test prior to starting therapy.
7. Female patients of childbearing potential and men must agree to use adequate contraception (at least one highly effective method and one additional method of birth control at the same time or complete abstinence) prior to study entry, for the duration of study participation and for at least 6 months following study drug discontinuation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. A female of childbearing potential (FCBP) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months (if age > 55 years); if the female subject is < 55 years and she has been naturally postmenopausal for > 1 year her reproductive status has to be verified by additional lab tests (< 20 estradiol OR estradiol < 40 with FSH > 40 in women not on estrogen replacement therapy).
8. Willingness and ability of the subject to comply with scheduled visits, drug administration plan, protocol specified laboratory tests, other study procedures, and study restrictions.
9. Evidence of a personally signed informed consent indicating that the subject is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation.

Exclusion Criteria:

1. Patients who have had prior radiotherapy to the head and neck region
2. Patients who are receiving any other investigational agents or an investigational device within 21 days before administration of first dose of study drugs.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to tolinapant.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
5. Significant cardiovascular disease (e.g., myocardial infarction, arterial thromboembolism, cerebrovascular thromboembolism) within 3 months prior to start of study therapy; angina requiring therapy; symptomatic peripheral vascular disease; New York Heart Association Class 3 or 4 congestive heart failure (or ejection fraction <50%); or uncontrolled Grade ≥3 hypertension (diastolic blood pressure ≥100 mmHg or systolic blood pressure ≥160 mmHg) despite antihypertensive therapy.
6. Contraindications to radiotherapy (e.g. uncontrolled connective tissue disorder).
7. Women who are pregnant or breast feeding.
8. Vulnerable populations including prisoners and adults who are unable to consent.
9. Known history of human immunodeficiency virus (HIV) infection, or seropositive results consistent with active hepatitis B virus (HBV) or active hepatitis C virus (HCV) infection.
10. Grade 3 or greater neuropathy.
11. Known distant metastases (i.e., outside of the neck).
12. Known significant mental illness or other conditions such as active alcohol or other substance abuse that, in the opinion of the investigator, predisposes the subject to high risk of noncompliance with the protocol treatment or assessments.
13. Concurrent second malignancy requiring active therapy.
14. Patients with a history of allogenic transplant must not have ≥Grade 3 graft-versus-host disease (GVHD) or any clinically significant GVHD requiring systemic immunosuppression.
15. Systemic corticosteroids >20 mg daily prednisone equivalent (unless patient has been taking a continuous dose for >3 weeks prior to study entry).
16. Medications known to cause QT prolongation including some antipsychotics (chlorpromazine, haloperidol, droperidol, quetiapine, olanzapine, amisulpride, thioridazine), antiarrhythmics (quinidine, procainamide, disopyramide, flecanide, encainide, sotalol, amiodarone), antidipressants (amitriptyline, doxepin, imipramine, nortriptyline, desipramine), mianserin, citalopram, escitalopram, venlafaxine, bupropion, moclobemide), and antihistamines (diphenhydramine, astemizole, loratadine, terfenadine), macrolide antibiotics (erythromycin, clarithromycin), and antimalarials (chloroquine, hydroxychloroquine, quinine), unless the use of these drugs cannot be avoided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2026-07-21 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole C Schmitt, MD, Principal Investigator — Emory University
Locations (1):
- Emory University/Winship Cancer Institute, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Tolinapant, Radiation Therapy)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Tolinapant, Radiation Therapy)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Safety of Tolinapant + Radiation (Number of Patients With Adverse Events Per CTCAE v5.0)
Description: Safety will be assessed on clinical examination and measurement of laboratory parameters. All safety assessments including adverse events, clinical laboratory evaluations, and vital signs will be summarized with descriptive statistics, where appropriate, and listed in the data listings using MedDRA terms.
Time Frame: Up to 60 days post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Tolinapant, Radiation Therapy)
Number analyzed (Participants) | 10
Participants | 10

2. Primary Outcome: Feasibility of Tolinapant + Radiation (Number of Patients Able to Complete Treatment)
Description: Feasibility is defined as completion of treatment, which will be reported as a percentage, with a 95% exact confidence interval using the Clopper-Pearson method.
Time Frame: Upon completion of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Tolinapant, Radiation Therapy)
Number analyzed (Participants) | 10
Participants | 10

ADVERSE EVENTS:
Time Frame: 2 years post treatment
Arm/Group | Treatment (Tolinapant, Radiation Therapy)
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Tolinapant, Radiation Therapy) (N=10)
Radiation Dermatitis (Skin and subcutaneous tissue disorders) | 10
Fatigue (General disorders) | 9
Anorexia (General disorders) | 9
Throat/Tumor Pain (Respiratory, thoracic and mediastinal disorders) | 8
Dysphagia (Respiratory, thoracic and mediastinal disorders) | 8
Dysgeusia (General disorders) | 7
Nausea (Metabolism and nutrition disorders) | 5
Dry Mouth (General disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-06): https://cdn.clinicaltrials.gov/large-docs/82/NCT05245682/Prot_SAP_000.pdf